CLINICAL TRIAL: NCT06862505
Title: Histological Analysis of Collagen Fibers Around Screw-less, Morse Taper Implant-abutment Connection 8 and 16 Weeks After Implant Uncovering: a Split-mouth Randomized Controlled Trial
Brief Title: Histological Analysis of Peri-implant Soft Tissue
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Università degli Studi di Sassari (Other)
Responsible Party: Principal Investigator, Marco Tallarico, Associate Professor, Università degli Studi di Sassari
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 15-16/12/24
Record Dates: First submitted 2025-02-25; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Implant Therapy; Biological Width
Keywords: Dental implants; Biological width; Istological analysis
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Biopsy at 8 weeks (Experimental)
  Interventions: Procedure: Biopsy
- Biopsy at 16 weeks (Active Comparator)
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — Biopsy of soft tissue were taken randomly at 8 or 16 weeks to compare soft tissue

SUMMARY:
The aim of this study is to evaluate the histologically analysis in humans and the orientation of collagen fibers around screw-less, morse taper implant-abutment connection.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older, affected by partial edentulism of posterior elements need for at least two single implant rehabilitations
* able to understand a sign an informed consent

Exclusion Criteria:

* Peapole having a systemic or local contraindications for implant placement;
* Untreated periodontal disease;
* smokers;
* osteoporosis;
* uncontrolled diabetes;
* refusal to implant rehabilitation;
* refusal to biopsy collection;
* systemic pathologies that could compromise the healing of peri-implant tissues.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
Histological analisys | 8 and 16 weeks
  Histological analysis of peri-implant gengivaat 8 and 16 weeks to assess collagen fibre orientation

SECONDARY OUTCOMES:
Histomorphometry | 8 and 16 weeks
  Quantitative measure of soft tissues

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rome, Rome, Italy, Italy

IPD SHARING:
Plan to Share IPD: No